CLINICAL TRIAL: NCT03495505
Title: Image Optimisation and Guidance for Wireless Endocardial Cardiac Resynchronisation Therapy: The CT Guided Trial
Brief Title: CT Guided WiSE-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 239322
Record Dates: First submitted 2018-03-26; First posted 2018-04-12 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
Keywords: WiSE-CRT; Endocardial Pacing Optimisation; Cardiac Resynchronisation Therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: 20 patients will be recruited into this feasibility study with a 6 month follow-up. There will be no blinding nor randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WiSE-CRT eligible (Experimental): Patients need to meet all the inclusion and none of the exclusion criteria in order to be eligible for the study. All these patients will receive the WiSE-CRT implant.
  Interventions: Device: WiSE-CRT

INTERVENTIONS:
Device: WiSE-CRT — Intervention will involve placement of the WISE-CRT system which consists of a transmitter, battery and electrode.
  Other Names: Cardiac Resynchronisation Therapy; Wireless Endocardial Pacing; WICS device

SUMMARY:
This feasibility study will use CT scanning to identify the optimal location for placement of the WiSE-CRT system.

DETAILED DESCRIPTION:
Heart failure (HF) is estimated to affect at least 10% of adults aged over 70 years old, with a 12-month all-cause mortality rate of 7% in stable patients. Cardiac resynchronisation therapy (CRT) is an important intervention for patients with severe left ventricular (LV) systolic impairment and helps to improve well-being and reduce morbidity and mortality. CRT is achieved by placing endocardial pacing leads into the right atrium and right ventricle and then placing a third pacing lead through the coronary sinus (CS) to enable epicardial LV pacing, thus achieving ventricular resynchronisation. Although this is a successful therapy, overall 30-40% of patients will fail to respond. Additionally, even in those eligible for CRT, approximately 8-10% of patients cannot have it implanted due to anatomical abnormalities such as venous occlusion, inappropriate CS targets, diffuse scar resulting in inappropriately high pacing thresholds or phrenic nerve stimulation. In these circumstances other avenues to achieve biventricular pacing needs to be sought.

The wireless CRT system (WiSE-CRT, EBR Systems) has been developed to overcome these issues. It uses an endocardial LV electrode to achieve biventricular pacing negating the need to implant a pacing lead through the CS. There are several advantages of endocardial LV pacing such as a greater selection of pacing sites, possibility of lower pacing outputs compared with conventional leads in the CS and it appears to be a more physiological way to pace. The WiSE-CRT system is used in conjunction with a single or dual-chamber pacemaker and is made up of several components. A transmitter is implanted subcutaneously, attached to a battery. This detects right ventricular pacing from the co-implant and then delivers ultrasonic energy which is received by an electrode placed in the LV endocardium to enable biventricular pacing. The transmitter must be placed in a position with an adequate "acoustic window," which requires a line from the transmitter to the LV that is free of significant tissue or bone. Additionally, the endocardial electrode must be placed in close proximity to the transmitter. In a study of 35 patients, the WiSE-CRT system was successful implanted in 97.1% of cases, with 97% achieving biventricular pacing at 1 month and 84.8% showing an improvement in the clinical composite score at 6 months. These results are particularly encouraging given the device was used in patients who had failed conventional CRT, representing a difficult patient group.

The major advantage of the WiSE-CRT system is that the LV electrode can be placed anywhere within the ventricle. Studies have shown that patient outcomes are improved by pacing at a site which avoids ventricular scar and targets an area of latest mechanical activation. These sites will vary according to the aetiology underlying HF. In addition, using conventional fluoroscopy to guide pacing lead implants has been shown to be inaccurate when compared with computed tomography (CT). Our group have previously shown that magnetic resonance imaging (MRI) can be overlaid on fluoroscopic images to help guide epicardial pacing to a specific location and improve outcomes. Many patients undergoing a WiSE-CRT implant will be unable to have a MRI due to their previous pacemaker implant. However, guidance may still be achieved using CT scanning.

The proximity and orientation of the transmitter to the endocardial electrode is important in determining the battery life of the WiSE-CRT system. Yeh et al. showed that a large proportion of patients have at least two suitable acoustic windows for placement of the transmitter. This provides the operator with more opportunities to carefully select an ideal location. However, once implanted the endocardial electrode must be placed within the acoustic window which limits the number of sites the electrode can then be placed.

Identifying the best location for both the transmitter and endocardial electrode is essential to target the most viable myocardium and improve patient outcomes. Ideally this should be achieved before the patient has undergone any procedure since implanting the transmitter limits the potential locations for the electrode. We believe CT guidance can provide satisfactory information to optimise the location for both the transmitter and electrode which will increase the patient response rate and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Ability to provide informed consent to participate and willing to comply with the clinical investigation plan and follow-up schedule.
* Patients with pre-existing permanent pacing systems in situ.
* Left ventricular systolic impairment with ejection fraction of <45%
* Clinical symptoms of heart failure despite optimal medical therapy (NYHA II- IV)
* QRS duration >120ms on surface ECG

Exclusion Criteria:

* Creatinine clearance <30mls/minute (GFR)
* Severe allergy to contrast medium or severe asthma/ COPD
* Life expectancy <1 year
* Significant aortic valve disease or prosthesis
* Significant mitral regurgitation
* Significant peripheral vascular disease
* Contraindication to anticoagulation therapy
* Insufficient acoustic window to the LV as assessed from diagnostic transthoracic echocardiography
* Left atrial or ventricular thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Change in acute haemodynamic response (dp/dt) during the procedure | Baseline and during procedure

SECONDARY OUTCOMES:
Change in Minnesota Living with Heart Failure Questionnaire Score | Baseline and 6 months
  This measures a change in the patients symptoms from baseline to 6-months post intervention. A higher value represents a better outcome.
Evidence of reverse remodelling (≥15% improvement in end systolic volume) on transthoracic echocardiogram at 6 months post CRT implantation | Baseline and 6 months
Change in 6 minute walk test | Baseline and 6 months
Change in cardio-pulmonary exercise test score | Baseline and 6 months
  This measures a change in the patients symptoms from baseline to 6-months post intervention. A higher value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Niederer, DPhil, Principal Investigator — King's College London
Locations (1):
- Guys and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Reddy VY, Miller MA, Neuzil P, Sogaard P, Butter C, Seifert M, Delnoy PP, van Erven L, Schalji M, Boersma LVA, Riahi S. Cardiac Resynchronization Therapy With Wireless Left Ventricular Endocardial Pacing: The SELECT-LV Study. J Am Coll Cardiol. 2017 May 2;69(17):2119-2129. doi: 10.1016/j.jacc.2017.02.059. PMID 28449772
- [Background] Ypenburg C, van Bommel RJ, Delgado V, Mollema SA, Bleeker GB, Boersma E, Schalij MJ, Bax JJ. Optimal left ventricular lead position predicts reverse remodeling and survival after cardiac resynchronization therapy. J Am Coll Cardiol. 2008 Oct 21;52(17):1402-9. doi: 10.1016/j.jacc.2008.06.046. PMID 18940531
- [Background] Miller MA, Neuzil P, Dukkipati SR, Reddy VY. Leadless Cardiac Pacemakers: Back to the Future. J Am Coll Cardiol. 2015 Sep 8;66(10):1179-89. doi: 10.1016/j.jacc.2015.06.1081. PMID 26337997